CLINICAL TRIAL: NCT02035163
Title: Atrial Fibrillation Prevention in Post Coronary Artery Bypass Graft Surgery With Cryoablation for Ganglionic Plexi
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, MD, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APIP
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Complication of Coronary Artery Bypass Graft; Atrial Fibrillation
Keywords: Atrial fibrillation; coronary artery bypass graft; cryoablation; ganglionic plexi
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Two sites cryoablation group (Active Comparator): Two ganglionic plexi around atrium was performed with 90-second cryoablation.
  Interventions: Procedure: Two sites cryoablation
- Control group (No Intervention): No Intervention group

INTERVENTIONS:
Procedure: Two sites cryoablation — Two ganglionic plexi around atrium was performed with 90-second cryoablation.
  Arms: Two sites cryoablation group

SUMMARY:
Atrial fibrillation after coronary artery bypass graft is a common complication.

The investigators have thought that the mechanism of temporarily postoperative atrial fibrillation is closely related to the autonomic nervous system imbalance.

In a last several years, cryoablation was substituted for atrial incision in many reports to simplify the maze procedure.

However, there has been no comparative study to delineate the feasibility of the use of cryoablation.

DETAILED DESCRIPTION:
Modified maze procedures that use energy sources for the ablation of atrial fibrillation concomitant with cardiac surgery have been shown to improve outcomes in patients with atrial fibrillation. Cryoablation of atrial fibrillation recently has been shown to lead to outcomes that were at least equivalent to those reported for other energy modalities over both short- and medium-term follow-up times.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery graft bypass patient
* sinus rhythm

Exclusion Criteria:

* Patients using antiarrhythmic
* severe hypotension after surgery ( systolic blood pressure <90mmHg)
* history of atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
freedom of atrial fibrillation or other atrial arrhythmia | 5 days after surgery
  check the occurrence of atrial fibrillation through EKG monitoring And bradycardia(<40/min) or tachycardia(>110/min) does not occur

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seog Oh, Ph.D, Study Chair — Seoul St. Mary's Hospital
Locations (1):
- The Catholic University of Korea, Seoul St Mary's Hospital, Seoul, Seo Cho Gu, South Korea

IPD SHARING:
Plan to Share IPD: No